CLINICAL TRIAL: NCT01452607
Title: A Phase 1, Double-blind, Placebo-controled, Randomized Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SPI-1005 (Ebselen)in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of SPI-1005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-101
Record Dates: First submitted 2011-10-10; First posted 2011-10-17 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Hearing Loss; Cancer
Keywords: Ebselen
MeSH Terms: conditions — Hearing Loss; Neoplasms | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SPI-1005 Capsule 200mg Ebselen x1 (Experimental): Lowest Dose Evaluated, 200mg Ebselen Total, Delivered as a Single Dose
  Interventions: Drug: SPI-1005
- SPI-1005 Capsule 200mg Ebselen x2 (Experimental): 2x Lowest Dose Evaluated, 400mg Ebselen Total, Delivered as a Single Dose
  Interventions: Drug: SPI-1005
- SPI-1005 Capsule 200mg Ebselen x4 (Experimental): 4x Lowest Dose Evaluated, 800mg Ebselen Total, Delivered as a Single Dose
  Interventions: Drug: SPI-1005
- SPI-1005 Capsule 200mg Ebselen x8 (Experimental): 8x Lowest Dose Evaluated, 1600mg Ebselen Total, Delivered as a Single Dose
  Interventions: Drug: SPI-1005
- SPI-1000 Capsule 0 mg Ebselen Placebo (Placebo Comparator): Matching Placebo Capsule, 0mg Ebselen Total, Delivered as a Single Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPI-1005 — 200 mg Ebselen oral capsules (SPI-1005), single dose
  Other Names: 200 mg Ebselen
  Arms: SPI-1005 Capsule 200mg Ebselen x1; SPI-1005 Capsule 200mg Ebselen x2; SPI-1005 Capsule 200mg Ebselen x4; SPI-1005 Capsule 200mg Ebselen x8
Drug: Placebo — 0 mg Ebselen oral capsules (SPI-1000), single dose
  Other Names: 0 mg Ebselen
  Arms: SPI-1000 Capsule 0 mg Ebselen Placebo

SUMMARY:
A study to determine the safety, tolerability, and pharmacokinetics of SPI-1005 capsules in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects
* Within 15% of their ideal weights (Table of "Desirable Weights of Adults," Metropolitan Life Insurance Company, 1983)
* Medically healthy subjects with clinically insignificant screening results (laboratory profiles, medical histories, ECGs, physical exam);
* Voluntarily consented to participate in the study;
* Females of childbearing potential were either sexually inactive (abstinent) for 14 days prior to screening and throughout the study or used one of the following acceptable birth control methods: Intrauterine device (IUD) in place for at least 3 months prior to study; Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; Stable hormonal contraceptive for at least 3 months prior to study through completion of study; Surgical sterilization (vasectomy) of partner at least 6 months prior to study. Females of non-childbearing potential were surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study, hysterectomy, or bilateral oophorectomy at least 2 months prior to study).

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, otologic, or psychiatric disease;
* History or presence of alcoholism or drug abuse within the past 2 years;
* Hypersensitivity or idiosyncratic reaction to compounds related to ebselen;
* Use of any prescription medication within 14 days (with the exception of hormonal contraceptives) prior to or during the study;
* Use of any over-the-counter medication including vitamins, herbal preparations, antacids, cough and cold remedies, etc., within 7 days prior or during the study;
* Use of any drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes within 28 days prior to dosing;
* Abnormal diet (for any reason) during the 30 days prior to dosing;
* Donation of whole blood within 56 days prior to the study;
* Plasma donation within 7 days prior to the study;
* Participation in another clinical trial within 30 days prior to the study;
* Female subjects who were pregnant or lactating;
* Hemoglobin < 12.0 g/dL;
* Orthostatic vital signs which result in: A pulse increase of more than 30 beats per minute after 3 minutes standing (compared with semi-recumbent pulse rate); or A pulse rate greater than 100 bpm after 3 minutes standing; or A drop in systolic blood pressure decrease of at least 20 mm Hg; or A diastolic blood pressure decrease of at least 10 mm Hg within 3 minutes of standing (compared with semi-recumbent blood pressure).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 month
  The primary objective of this study was to evaluate the safety and tolerability of SPI-1005 (ebselen) in healthy subjects. Incidence and severity of Adverse Events were determined in all treatment and placebo groups.

SECONDARY OUTCOMES:
Pharmacokinetics of SPI-1005 and its major metabolites in healthy subjects | 24 hours
  Evaluate the single dose pharmacokinetic profile of SPI-1005 in healthy subjects including Tmax, Cmax, of the parent compound and major metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Kisicki, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lynch E, Kil J. Development of Ebselen, a Glutathione Peroxidase Mimic, for the Prevention and Treatment of Noise-Induced Hearing Loss. Semin Hear 2009; 30(1): 047-055
- [Derived] Garland M, Hryckowian AJ, Tholen M, Bender KO, Van Treuren WW, Loscher S, Sonnenburg JL, Bogyo M. The Clinical Drug Ebselen Attenuates Inflammation and Promotes Microbiome Recovery in Mice after Antibiotic Treatment for CDI. Cell Rep Med. 2020 Apr 21;1(1):100005. doi: 10.1016/j.xcrm.2020.100005. PMID 32483557